CLINICAL TRIAL: NCT00685412
Title: Phase I Open Label, Dose Escalation Study to Evaluate the Safety, Tolerability and Immunogenicity of Human Papillomavirus (HPV) DNA Plasmid (VGX-3100) + Electroporation (EP) in Adult Females Post Surgical or Ablative Treatment of Grade 2 or 3 Cervical Intraepithelial Neoplasia (CIN)
Brief Title: Phase I of Human Papillomavirus (HPV) DNA Plasmid (VGX-3100) + Electroporation for CIN 2 or 3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HPV001
Record Dates: First submitted 2008-05-22; First posted 2008-05-28 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Papillomavirus Infections
Keywords: CIN 2 or 3; cervical cancer
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms | interventions — VGX-3100

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0.6mg of DNA/dose (Experimental): Subjects will receive a 3 dose series of VGX-3100 containing 0.6mg DNA/dose administered via IM injection + electroporation at Day 0, Month 1 and Month 3
  Interventions: Biological: VGX-3100
- 2mg of DNA/dose (Experimental): Subjects will receive a 3 dose series of VGX-3100 containing 2mg of DNA/dose administered via IM injection + electroporation at Day 0, Month 1 and Month 3
  Interventions: Biological: VGX-3100
- 6mg of DNA/dose (Experimental): Subjects will receive a 3 dose series of VGX-3100 containing 6mg DNA/dose administered via IM injection + electroporation at Day 0, Month 1 and Month 3
  Interventions: Biological: VGX-3100

INTERVENTIONS:
Biological: VGX-3100 — DNA plasmid delivered via IM injection + electroporation using CELLECTRA device

SUMMARY:
DNA vaccines, which are small pieces of DNA also known as plasmids, have several advantages over traditional vaccines such as live attenuated virus and recombinant protein-based vaccines. DNA vaccines appear to be well tolerated in humans. Therefore, we have developed our DNA vaccine, VGX-3100, to include plasmids targeting E6 and E7 proteins of both HPV subtypes 16 and 18. We have chosen to deliver our candidate vaccines via electroporation (EP) using the CELLECTRA™ constant current device to deliver a small electric charge following intramuscular (IM) injection, since animal studies have shown that this delivery method increases the immune response to our DNA vaccine leading to a decrease in the size of tumors caused by HPV 16 and 18. The vaccine is proposed to be given to patients with a history of CIN 2 and 3 that have been treated by surgery. We will determine which dose the DNA vaccine will be the best tolerated and elicit the strongest immune response.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent in accordance with institutional guidelines;
* Female 18-45 years of age;
* Post surgical (including LEEP and conization) or ablative treatment and a diagnosis of CIN 2 or 3, while under physician care as per ASCCP guidelines (Appendix D);
* Normal ECG and normal laboratory values as judged by Grade 0-1 as per Toxicity Grading Scale for Healthy Adults (Appendix C) for CBC, CPK, SMA-12 and urinalysis evaluations done up to 30 days prior to administration of study treatment;
* Body mass index (BMI) ≤30 kg/m2;
* Women of child-bearing potential (WOCBP) agree to remain sexually abstinent, use medically effective contraception (oral contraception, barrier methods, spermicide, etc), or have a partner who is sterile (i.e., vasectomy) from enrollment to 3 months after the last injection (~6 months);
* Able and willing to comply with all study procedures.

Exclusion Criteria:

* Active infection with herpes simplex virus (HSV);
* Positive serological test for HIV virus, hepatitis C virus or Hepatitis B virus surface antigen (HBsAg);
* Pregnant or breastfeeding subjects;
* Any concurrent condition requiring the continued use of systemic or topical steroids (excluding inhaled and eye drop-containing corticosteroids) or the use of immunosuppressive agents. All other corticosteroids must be discontinued > 4 weeks prior to Day 1 of treatment;;
* Administration of any blood product within 3 months of enrollment;
* Administration of any vaccine within 6 weeks of enrollment;
* Patient is currently participating or has participated in a study with an investigational compound or device within 30 days of signing informed consent;
* Metal implants at the site of injection;
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements;
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (i.e. infections disease) illness must not be enrolled into this study;
* Any other conditions judged by the investigator that would limit the evaluation of a subject.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-05; Primary Completion 2011-01 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of escalating doses of VGX-3100, administered by IM injection with EP to adult female subjects post surgical or ablative treatment of grade 2 or 3 CIN. | Through Month 4

SECONDARY OUTCOMES:
Humoral and cellular immune responses to VGX-3100 in blood samples obtained from study subjects after each dose of a 3-dose series of VGX-3100 containing 0.6, 2 or 6 mg of DNA/dose. | At end of study

CONTACTS AND LOCATIONS:
Overall Officials: Christina Chu, MD, Principal Investigator — University of Pennsylvania; Robert Parker, MD, Principal Investigator — Lyndhurst Gynecologic Associates; John Sunyecz, MD, Principal Investigator — Laurel Highlands, OB/GYN, P.C.; Javier Morales, MD, Principal Investigator — Clinical Research Puerto Rico
Locations (4):
- United States (3):
  - Lyndhurst Gynecologic Associates, Winston-Salem, North Carolina
  - Laurel Highlands, OB/GYN, P.C., Hopwood, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
- Clinical Research Puerto Rico, San Juan, Puerto Rico